CLINICAL TRIAL: NCT00902811
Title: Comparing the Effectiveness of 5 Artemisinin Combination Treatment Regimens in the Treatment of Uncomplicated Falciparum Malaria
Brief Title: Effectiveness of Artemisinin Combination Regimens in Falciparum Malaria
Acronym: ACT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Collaborators: Mahidol University (Other); University of Oxford (Other); Disease Control, Department of Health, Myanmar (Unknown)
Responsible Party: Frank Smithuis, Medecins Sans Frontieres, Holland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YNG0901
Record Dates: First submitted 2009-04-30; First posted 2009-05-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Uncomplicated Falciparum Malaria
Keywords: uncomplicated falciparum malaria; artemisinin combination therapy
MeSH Terms: interventions — Mefloquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- AM(LT) (Active Comparator): Artesunate (Arsumax®, Sanofi)
  Interventions: Drug: AM(LT)
- AM(FDC) (Experimental): Artesunate-mefloquine fixed dose combination
  Interventions: Drug: AM(FDC)
- AL (Experimental): artemether 20 mg - lumefantrine 120 mg co-formulated tabs
  Interventions: Drug: AL
- DP (Experimental): 40 mg dihydroartemisinin/320 mg piperaquine tablets and Dihydropiperaquine 20mg/Piperaquine 160 mg tablets
  Interventions: Drug: DP
- AA (FDC) (Experimental): Artesunate-amodiaquine fixed dose combination
  Interventions: Drug: AA(FDC)

INTERVENTIONS:
Drug: AM(FDC) — Artesunate-mefloquine fixed dose combination (artesunate 25mg/mefloquine hydrochloride 55mg, or artesunate 100mg/mefloquine hydrochloride 220mg), according to age-group.
  Other Names: Far-Manguinhos, Brazil
  Arms: AM(FDC)
Drug: AM(LT) — Artesunate (Arsumax®, Sanofi) 50 mg tabs given at 4 mg/Kg/day on day 0, day 1 and day 2 (total 12 mg/Kg) PLUS Mefloquine 250 mg base tabs given at 25 mg/Kg on day 0. Treatment is given in three equally divided daily doses to the nearest quarter tablet.
  Other Names: Lariam®, Roche
  Arms: AM(LT)
Drug: AL — Coartem®: artemether 20 mg - lumefantrine 120 mg co-formulated tabs (Coartem®, Novartis) given as six twice-daily doses over three days, according to weight-groups. The second dose should be taken 6 to 10 hours after the first dose, given at inclusion. Patients will be advised to take some fatty food (or encouraged to give breast feeding) before each dose is taken. Fatty food or milk will not be provided by the researchers.
  Other Names: Coartem®
  Arms: AL
Drug: DP — 40 mg dihydroartemisinin/320 mg piperaquine tablets and Dihydropiperaquine 20mg/ Piperaquine 160 mg tablets),. Treatment is given according to age groups. In the age group <6yrs of age, a subdivision according to weight is made
  Other Names: DuoCotecxin, Holley Pharm
  Arms: DP
Drug: AA(FDC) — Artesunate-amodiaquine fixed dose combination (FDC) (Artesunate Amodiaquine Winthrop® Sanofi Aventis); Artesunate 25mg/amodiaquine 67.5mg; Artesunate 50mg/amodiaquine 135mg ; Artesunate 100mg/amodiaquine 270mg
  Other Names: Artesunate Amodiaquine Winthrop® Sanofi Aventis
  Arms: AA (FDC)

SUMMARY:
Antimalarial drug resistance is increasing nearly everywhere in the tropical world, confounding global attempts to "Roll Back Malaria." South East Asia has the most resistant malaria parasites in the world. This has limited the options for treatment in this region.

Artemisinin-based combination therapy is now the recommended treatment for uncomplicated falciparum malaria. The success of this policy change in practice will depend on the efficacy of the components of the combination used, the population coverage achieved, high levels of adherence to treatment, low cost of the drugs, and preferably the drugs in a combination treatment should be formulated in a single tablet, to prevent one drug being taken without the partner drug. Until recently there were only two artemisinin-based fixed combinations available, artemether-lumefantrine and dihydroartemisinin-piperaquine; and only the former has international registration. More fixed combinations are needed urgently.

DETAILED DESCRIPTION:
Malaria in Myanmar:

In Myanmar, malaria is the number one cause of morbidity. According to the Department of Health (DoH) and WHO there are approximately 500,000 patients with malaria each year. About 80% of reported infections are due to Plasmodium falciparum and 20% are due to Plasmodium vivax. This is likely to be a severe underestimation. MSF-Holland alone treats already 250,000 slide positive malaria patients per year in an area of mixed endemicity covering a population of less that 1 million patients out of a total population of 54 million in the country.

Chloroquine was the first line treatment for falciparum malaria for the last five decades. In 1996 and 1998 MSF-Holland with support from the Wellcome Trust (Prof N. White) performed studies in the northern and western part of the country, in which very high in-vivo resistance levels to chloroquine and sulfadoxine-pyrimethamine were demonstrated1,2. Combination treatment of mefloquine plus artesunate (loose tablets) [MA(LT)]and treatment with dihydroartemisinin-piperaquine (DP) both proved highly efficacious (99-100%)3,4. The studies performed by MSF provided an important component of the evidence used to convince the health authorities that a change of national protocol was needed. In 2001, the DOH of Myanmar changed the national protocol for the treatment of uncomplicated falciparum malaria; a 3 day treatment of mefloquine-artesunate was chosen to become the first line treatment. Artemether-lumefantrine (AL) and DP are also mentioned in the national protocol as effective treatment regimens, but there is a call in the protocol for more research of these treatments.

These changes in policy are a very good step forward and were widely respected. In practice, some problems remain.

MSF has implemented large malaria activities in Myanmar over the past decade. The programme has performed a diagnostic test for malaria for approximately 3,000,000 patients and approximately 1,500,000 patients have been treated with artemisinin combination treatment (ACT).

ELIGIBILITY:
Inclusion criteria

* Age over 6 months and
* Weight ≥ 5 kg, and
* Slide-confirmed infection with Plasmodium falciparum (including mixed infections), and
* Asexual parasite density between 500 and 200,000/µl of blood, and
* Informed consent from a parent or guardian aged at least 18 years.

Exclusion criteria

* General danger signs according to the WHO definition or
* Signs of severe/complicated malaria according to the WHO definition or
* Severe anaemia (haemoglobin < 5 g/dL), or
* Known history of hypersensitivity to any of the study drugs, or
* Severe malnutrition (as defined by a weight-for-height below 70% of median and/or symmetrical oedemas involving at least the feet), or
* Concomitant febrile illness due to causes other than malaria with the potential to confound study outcome (measles, acute lower tract respiratory infection, otitis media, tonsillitis, abscesses, severe diarrhoea with dehydration, etc.; mild flu should not lead to exclusion) or
* History of psychiatric diseases, or
* Having received a full course treatment including MQ in the preceding 9 weeks or
* Having received any other antimalarials in the previous 48 hours.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 63 days

SECONDARY OUTCOMES:
Early treatment failure | Day 6
Late treatment failure | Day 63
Adequate response | Day 63

CONTACTS AND LOCATIONS:
Overall Officials: Frank Smithuis, MD, Principal Investigator — Medecins Sans Frontieres, Netherlands
Locations (4):
- Burma (4):
  - Dabhine and Mingan Clinic, Sittwe, Rakhine State
  - Myit Kyi Nar Clinic, Kachin
  - Myothugyi Rural Health Center, Bu Thee Daung, Maungdaw
  - Lashio Clinic, Shan

REFERENCES:
- [Derived] Smithuis F, Kyaw MK, Phe O, Win T, Aung PP, Oo AP, Naing AL, Nyo MY, Myint NZ, Imwong M, Ashley E, Lee SJ, White NJ. Effectiveness of five artemisinin combination regimens with or without primaquine in uncomplicated falciparum malaria: an open-label randomised trial. Lancet Infect Dis. 2010 Oct;10(10):673-81. doi: 10.1016/S1473-3099(10)70187-0. Epub 2010 Sep 9. PMID 20832366